CLINICAL TRIAL: NCT06338202
Title: Real-World Effectiveness of MAVacamtEN in Canada (MAVEN): A Retrospective Physician Survey of Patient Charts
Brief Title: Real-World Effectiveness of Mavacamten in Canada
Acronym: MAVEN
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV027-1137
Record Dates: First submitted 2024-03-25; First posted 2024-03-29 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy (oHCM)
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with mavacamten: Patients with symptomatic obstructive hypertrophic cardiomyopathy (NYHA functional class II-III) who receive mavacamten as part of routine clinical care
  Interventions: Drug: Mavacamten

INTERVENTIONS:
Drug: Mavacamten — As detailed in the product label

SUMMARY:
The purpose of this observational, retrospective, physician survey study is to describe the real-world effectiveness and use of mavacamten in participants who initiated treatment for obstructive hypertrophic cardiomyopathy (oHCM) in Canada.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have initiated mavacamten, as part of routine clinical care, through the Bristol Myers Squibb CAMZYOS Patient Support Program for the treatment of symptomatic obstructive hypertrophic cardiomyopathy (oHCM)
* Adult patient (≥18 years of age or as defined per local province/territory) at Index Date (first prescribed dose of mavacamten).
* Patient has been diagnosed with symptomatic oHCM of New York Heart Association (NYHA) class II to III at the time of mavacamten initiation.

Exclusion Criteria:

* In the 6 weeks prior to baseline (i.e., Index Date; date of first prescribed dose of mavacamten), patient has received any cardiac myosin inhibitor (including mavacamten) for oHCM or any other medical condition as part of a clinical trial.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The observational study will include adult patients with symptomatic obstructive hypertrophic cardiomyopathy (oHCM) who are enrolled in the Bristol Myers Squibb (BMS)-sponsored CAMZYOS Patient Support Program and who have initiated mavacamten as part of routine clinical care in Canada.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Change in New York Heart Association (NYHA) functional class following mavacamten treatment initiation | Up to 1.5 years
  * Proportion of patients in each New York Heart Association (NYHA) functional class following mavacamten treatment initiation
  * Proportion of patients with a reduction of ≥1 New York Heart Association (NYHA) functional class following mavacamten treatment initiation

SECONDARY OUTCOMES:
Change in left ventricular outflow tract (LVOT) with Valsalva maneuver (vLVOT) gradient following mavacamten treatment initiation | Up to 1.5 years
Proportion of patients with left ventricular outflow tract (LVOT) with Valsalva maneuver gradient (vLVOT) < 20mmHg following mavacamten treatment initiation | Up to 1.5 years
Age | Baseline
Sex at birth | Baseline
Ethnicity | Baseline
Employment status | Baseline
Body mass index (BMI) | Baseline
Obstructive hypertrophic cardiomyopathy (oHCM) disease duration | Baseline
Proportion of patients in each New York Heart Association (NYHA) functional class II and III | Baseline
Left ventricular outflow tract (LVOT) with Valsalva maneuver (vLVOT) gradient | Baseline
Left ventricular ejection fraction by 2D echocardiogram (LVEFb) | Baseline
Mavacamten dose regimen | Up to 1.5 years
Proportion of patients who discontinued mavacamten | Up to 1.5 years
Duration of treatment prior to mavacamten discontinuation | Up to 1.5 years
Left ventricular ejection fraction by 2D echocardiogram (LVEF) at the time of mavacamten treatment discontinuation | Up to 1.5 years
Proportion of patients with left ventricular ejection fraction by 2D echocardiogram (LVEF) < 50% at the time of mavacamten treatment discontinuation | Up to 1.5 years
Reason for discontinuing mavacamten treatment | Up to 1.5 years
Functional assessment schedule | Up to 1.5 years
  * Proportion of patients who undergo left ventricular outflow tract with Valsalva maneuver gradient (vLVOT) functional assessment
  * Proportion of patients who undergo left ventricular ejection fraction (LVEF) assessment

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- London Health Science Centre (LHSC), London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts